CLINICAL TRIAL: NCT05274048
Title: A Multi-Center Phase I Trial of Neratinib and Fam-trastuzumab Deruxtecan in Advanced Refractory Gastric and Esophageal Cancer Patients
Brief Title: Neratinib and Fam-Trastuzumab Deruxtecan in Advanced Gastro-esophageal Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-1069; GI-200 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2022-01-28; First posted 2022-03-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Gastric Cancer; Gastrointestinal Cancer; HER2 Gene Mutation
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neratinib plus TDxD (Experimental): Neratinib oral daily days 1-21 plus TDxD on day 1 administered intravenously of a 21 day treatment cycle.
  Interventions: Drug: Neratinib Pill; Drug: Fam-Trastuzumab Deruxtecan-Nxki (TDxD)

INTERVENTIONS:
Drug: Neratinib Pill — Patients will be enrolled in cohorts of 3 at each dose level of Neratinib (120 mg, 160 mg, 200 mg) daily (days 1 through 21)
Drug: Fam-Trastuzumab Deruxtecan-Nxki (TDxD) — standard dosing of TDxD (5.4mg/m2) on day 1of a 21 day treatment cycle

SUMMARY:
This is Phase 1 dose finding trial with potential dose expansion to evaluate the safety, toxicity, recommended phase 2 dose (RP2D), and maximum tolerated dose (MTD) of Neratinib plus TDxD using a standard 3+3 dose escalation design in patients with metastatic or unresectable gastro-esophageal cancer that are HER2-overexpressing (IHC 3+ or IHC2+/ISH+) and any other gastrointestinal cancer with HER2 expression with IHC3+. Patients must have progressed or been intolerant of at least one prior line of chemotherapy + HER2 directed therapy.

DETAILED DESCRIPTION:
This is Phase 1 dose finding trial with potential dose expansion to evaluate the safety, toxicity, recommended phase 2 dose (RP2D), and maximum tolerated dose (MTD) of Neratinib plus TDxD using a standard 3+3 dose escalation design in patients with metastatic or unresectable gastro-esophageal cancer that are HER2-overexpressing (IHC 3+ or IHC2+/ISH+) and any other gastrointestinal cancer with HER2 expression with IHC3+. Patients must have progressed or been intolerant of at least one prior line of chemotherapy + HER2 directed therapy. A total of 18 patients will be enrolled with the plan to reach MTD and enroll any remaining patients at the RP2D to further define the toxicities and preliminary efficacy to help define the future studies with this combination. Patients will be enrolled in cohorts of 3 at each dose level (see SCHEMA). It is anticipated that the trials may escalate through 3 different dose levels of Neratinib (120 mg, 160 mg, 200 mg) and standardized approved dosing of TDxD (5.4mg/kg) in breast cancer will be used as explained in the study rationale. Both drugs have GI toxicity specifically diarrhea and the combination may have risk of increased toxicity from TDxD due to increase cellular uptake of the cytotoxic payload. Therefore, we are not testing the recommended single agent dose of 240mg of Neratinib with this combination. For the same reason, TDxD will not be used at the approved single agent dose of 6.4mg/kg as the safety of this dosing was established in the monotherapy setting [33]. If the initial dose level 0 is deemed too toxic, the study investigators and DSMB can make a decision to allow dose reduction of TDxD to 4.4mg/kg (dose level -1) and reintroduction of neratinib at dose level 0, if the toxicities are felt to be related to TDxD. For cycle 1, patients will start with Neratinib lead in starting at Day -7 and TDxD will be administered on Day 1. Each future treatment cycle will comprise of Neratinib administered PO daily for a 21-day cycle with food. TDxD will be administered intravenously on day 1 of a 21-day cycle. The Dose Limiting Toxicities (DLT) window to determine MTD for the trial will be 28 days (cycle 1) from the start of the treatment. If toxicities are experienced outside the DLT window, they would not be considered in determining the MTD but will be closely monitored by the study team as well as institutional DSMB to ensure patient safety. The 28-day window will also help determine the RP2D. At the conclusion of the safety lead in portion, the Cohort Review committee will determine the RP2D, based on MTD as well as the safety profile of the drug after careful consideration. DLT will be defined in this study as a clinically significant adverse event or abnormal laboratory value assessed as described in section 6.3. All patients will undergo screening transthoracic echocardiography or multigated acquisition scan (MUGA) prior to initiating treatment and every 12 weeks while on treatment. The same imaging tumor assessment as at the time of screening should be used (computed tomography (CT) of the chest abdomen and pelvis with IV contrast or CT of the chest without IV contrast and magnetic resonance imaging (MRI) of the abdomen/pelvis if iodinated contrast is contraindicated). Tumor assessment must be performed every 3 cycles (+/-7 days). The assessment will be conducted before day 1 of each cycle as possible. Head CT/MRI should only be done when symptoms associated with brain metastasis occur.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have been diagnosed with histologically or cytologically confirmed gastrointestinal cancer (esophagus, stomach, colon, biliary, pancreas or unknown primary likely GI), and been deemed unresectable or have at least one site of metastatic disease
2. Patients must have evaluable or measurable disease by RECIST 1.1 criteria
3. 4.1.3 Patients' tumors must have HER2-overexpressing:

   1. (IHC 3+ or IHC2+/ISH+) advanced gastroesophageal cancer (including gastroesophageal junction adenocarcinoma).
   2. IHC 3+ for other GI cancers
4. Patients must have received at least one prior line of HER2 directed therapy for metastatic/unresectable disease and completed treatment at least 2 weeks prior to C1D1 (only for Gastroesohageal cancers, not for other GI cancers)
5. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
6. Age > 18 years.
7. ECOG performance status 0-2
8. Patients must have normal organ and marrow function as defined below

   * Leukocytes > 3,000/mcL
   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 90,000/mcL
   * Hemoglobin > 9 gm/dl
   * Total bilirubin < 2 times institutional normal limits
   * AST/ALT (SGOT/SGPT) < 5 times institutional normal limits if liver metastases and </+ 2 times institutional normal limits otherwise
   * Creatinine < 2.0mg/dL OR
   * Creatinine clearance > 50 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal
9. Left Ventricular Ejection Fraction ≥ 45% or lower limit of normal.
10. Chemotherapy is harmful to the human fetus. For this reason, females of childbearing potential must be willing to use an effective method of contraception, as outlined in Section 4.4, for the course of the study through at least 6 months after the last dose of study medication. Males who have women of childbearing (WOCB) partners must agree to use an effective method of contraception as outlined in Section 4.4 for the course of the study through 8 months after the last dose of study medication.
11. Patients should be willing and able to swallow oral tablet medications
12. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Patients who have had chemotherapy, or radiotherapy within 2 weeks prior to C1D1 or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier (secondary hypothyroidism from prior immunotherapy is permissible if controlled on thyroid hormone replacement). Recovery is defined as any treatment onset adverse events returning to baseline or otherwise deemed not clinically significant.
2. Patients may not be receiving any other investigational agents for advanced cancer and must not have received prior treatment with TDxD
3. Immunotherapy and treatments involving any investigational agents must be discontinued for >21 days before Cycle 1 Day 1 (C1D1)
4. Patients with known untreated brain metastases are excluded from this study because of their poor prognosis and frequent development of neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Treated brain metastases are allowed (requires stability on MRI at least 4 weeks after initial treatment). Patients with treated brain metastases are allowed to be treated with steroid and/or anti-convulsants if the dose remains stable or decreases over the last 4 weeks prior to C1D1
5. Patients with ongoing diarrhea (> 4 bowel movements/day) unresolved despite medical and best supportive care in the two weeks preceding therapy
6. Patients will be excluded if they have had interstitial lung disease or pneumonitis or were suspected to have interstitial lung disease or pneumonitis that could not be ruled out on imaging at screening or if they had a history of noninfectious interstitial lung disease or pneumonitis that had been treated with glucocorticoids. Similarly, patients with clinically significant lung disease requiring O2 support or impaired lung function per investigator should be excluded
7. History of allergic reactions attributed to compound of similar chemical or biologic composition to the agent(s) used in this study
8. Patients receiving any medications or substances that are strong inhibitors or inducers of Neratinib and/or TDxD are ineligible.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Has a QT interval corrected by Fridericia's formula (QTcF) prolongation to >470 msec (female subjects) or >450 msec (male subjects) based on average of the Screening triplicate12-lead ECG.
11. Any patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, including uncontrolled HIV with CD4 count <200, untreated Hepatitis B are excluded from the study. Patients who have been treated for hepatitis C definitively with evidence of sustained virologic response, as well as HIV and hepatitis B patients on treatment with undetectable viral load will be eligible for inclusion.
12. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of the combination of TDxD and Neratinib | 2 years
  The rate of dose-limiting toxicities (DLTs) for Neratinib + TDxD during DLT period of 28 days, in patients with advanced gastrointestinal cancer

SECONDARY OUTCOMES:
Determine the Objective Response Rate (ORR) (Complete Response (CR) + Partial Response (PR)) of the combination of TDxD and Neratinib | 2 years
  Rate of grade 3 or higher adverse events with TDxD and Neratinib in patients with advanced gastrointestinal cancer
Determine the Disease Control Rate (DCR) (CR + PR + Stable Disease (SD)) of the combination of TDxD and Neratinib | 2 years
  Objective Response Rate (ORR) of the combination of TDxD and Neratinib in patients with advanced gastrointestinal cancer (Complete and partial response per RECIST 1.1)
Determine the Progression Free Survival (PFS) of the combination of TDxD and Neratinib | 2 years
  Progression Free Survival (PFS) of the combination of TDxD and Neratinib in patients with advanced gastrointestinal cancer (time from treatment initiation to disease progression or death from any cause)
Determine the Overall Survival (OS) of the combination of TDxD and Neratinib | 2 years
  Overall Survival (OS) of the combination of TDxD and Neratinib in patients with advanced gastrointestinal cancer (defined as the time from treatment initiation to death from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Namrata Vijavergia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Stanford Cancer Center, Palo Alto, California
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No